CLINICAL TRIAL: NCT06257095
Title: Improving Adult Protective Services Client Outcomes: A Stepped-Care Social and Mental Health Engagement Program
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Collaborators: Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Principal Investigator, Jason Burnett, Associate Professor, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: HSC-MS-23-0344
Record Dates: First submitted 2024-02-05; First posted 2024-02-13 (Actual); Last update posted 2024-02-13 (Actual); Status verified 2024-02

CONDITIONS: Depression in Old Age
Keywords: social engagement; Adult Protective Services (APS); elder abuse; self neglect

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Treatment (Experimental)
  Interventions: Behavioral: Stepped-care social and mental health engagement; Behavioral: APS Usual care
- Usual Care (Active Comparator)
  Interventions: Behavioral: APS Usual care

INTERVENTIONS:
Behavioral: Stepped-care social and mental health engagement — Each student will be matched to an older adult and the students will make one call o the older adult which lasts upto 1 hour each week for 8 weeks. Ending each call, the student will assess symptoms of depression anxiety through questionnaires. If the participant responds yes on two consecutive calls to any of these questions, they will be asked if they would like to receive a call from the University of Texas Health Science Center Trauma and Resilience Center to discuss free counseling services.
  Arms: Treatment
Behavioral: APS Usual care — Participants will receive a phone call for data collection. Then they will be offered to receive an abbreviated version of the stepped-care social and mental health engagement intervention, lasting only 6-weeks with the option to continue calls if agreeable between the student and older adult.

SUMMARY:
The purpose of this study is to ascertain the feasibility and effectiveness of an 8-week social engagement program aimed at reducing depression and increasing social engagement among seniors who are transitioning out of Adult Protective Services (APS) for either elder abuse or self-neglect.

ELIGIBILITY:
Inclusion Criteria:

Older Adults

* an APS validated EM/SN case
* able to provide informed consent
* able to speaks English or Spanish,
* community-dwelling,
* able to hear sufficiently using the telephone
* transitioning out of APS intervention (i.e. in the case closure phase of the APS service).

Student

* college or university student
* enrolled at one of the UTHealth graduate programs in Houston, University of Houston, Texas Southern University, Sam Houston State University, or Rice University
* commit to making 8-weekly consecutive calls
* complete the required 1-hour training and assessment.

Exclusion Criteria:

Older Adults

* Individuals needing a proxy to consent
* suspected or confirmed decision-making capacity impairments or uncontrolled psychiatric illnesses such as schizophrenia, paranoia, delusion, or delirium
* Older adults transitioning to a nursing home, assisted-living, or residential care facility

Student

-only engaging in the program to fulfill some educational requirement

Min Age: 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2023-08-09 (Actual); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-06-01 (Estimated)

PRIMARY OUTCOMES:
Change in social isolation assessed by the Duke Social Support Index (DSSI-6) | baseline, 4-week and 8-week follow-up
  This is a 6-item questionnaire and each is measured from 1(hardly ever) to 3(most of the time) for a maximum score of 18, higher score indicating greater social support
Change in loneliness as assessed by the University of California Los Angeles (UCLA )loneliness scale | baseline, 4-week and 8-week follow-up
  This is a 20-item questionnaire , each item is rated as either O ("I often feel this way"), S ("I sometimes feel this way"), R ("I rarely feel this way"), N ("I never feel this way") for a score range of 0-3,for a maximum score of 60, higher score indicating worse outcome
Change in depression as assessed by the PATIENT HEALTH QUESTIONNAIRE (PHQ-9) | baseline, 4-week and 8-week follow-up
  This is a 9 item questionnaire and each is scored from 0(not at all) to 3(nearly every day) , for a maximum score of 27 , higher score indicating more depression
Recurrence of Elder mistreatment (EM) | From participant's first call to 1 month post final call
  This is a yes or no questionnaire that will be answered by adult protective services (APS)
Recurrence of self neglect (SN) | From participant's first call to 1 month post final call
  This is a yes or no questionnaire that will be answered by adult protective services (APS)

SECONDARY OUTCOMES:
Change in anxiety as assessed by the Generalized Anxiety Disorder scale (GAD-7) | baseline, 4-week and 8-week follow-up
  This is a 7-item questionnaire , each is scored from 0(not at all) to 3(nearly every day), for a score range of 0-21 higher score indicating more anxiety
Change in resilience as assessed by the Brief Resilience Scale | baseline, 4-week and 8-week follow-up
  This is a 6-item questionnaire, questions 1, and 5 are scored from 1(strongly disagree) to 5(strongly agree) and questions 2, 4 and 6 are reverse scored , for a score range of 6-30. The total score is then divided by the number of questions answered to get the final score. higher score indicating more resilience.

CONTACTS AND LOCATIONS:
Overall Officials: Jason Burnett, PhD, Principal Investigator — The University of Texas Health Science Center, Houston
Locations (1):
- The University of Texas Health Science Center at Houston, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No